CLINICAL TRIAL: NCT07331597
Title: Effects of Scapulothoracic Joint Mobilization With or Without Acromioclavicular Joint Mobilization in Patients With Sub-acromial Pain Syndrome
Brief Title: Scapulothoracic Joint Mobilization With or Without Acromioclavicular Joint Mobilization in Sub-acromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0185
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sub-acromial Pain Syndrome
Keywords: soulder pain, scapulothoracic joint mobilization, acromioclavicular joint mobilization, sub-acromial pain syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Scapulothoracic joint mobilization with acromioclavicular joint mobilization
  Interventions: Other: Scapulothoracic joint mobilization; Other: Acromioclavicular joint mobilization; Other: Standard physiotherapy treatment
- Group B (Active Comparator): Scapulothoracic joint mobilization
  Interventions: Other: Scapulothoracic joint mobilization; Other: Standard physiotherapy treatment

INTERVENTIONS:
Other: Scapulothoracic joint mobilization — during 1st week of treatment, patients received Maitland grade-II mobilization for upward rotation, posterior tilting and external rotation glide, 5-10 oscillations per minute, 3 sets with 10 repetitions with 30 seconds rest interval. during 2nd, 3rd and 4rth week, patients received grade- II and III Maitland mobilization for upward rotation, posterior tilting and external rotation glide, 3 sessions a week for 4 weeks
Other: Acromioclavicular joint mobilization — during 1st week : Maitland grade-II mobilization for AC joint inferior glide, 5-10 oscillations per minute, 3 sets with 10 repetitions with 30 seconds rest interval. during 2nd, 3rd and 4rth week : Maitland grade-II, III for AC joint inferior glide, 5-10 oscillations per minute, 3 sets with 10 repetitions with 30 seconds rest interval, 3 sessions a week for 4 weeks.
  Arms: Group A
Other: Standard physiotherapy treatment — Moist hot pack for 10-15 minutes on shoulder region in supine lying position. TENS modulated mode for 10 minutes. Scapular stabilization exercises including: scapular protraction and retraction, shoulder extension, shoulder external rotation, standing snow angels, standing weight shift, ball stabilization exercise, serratus anterior punch. 3 sets with 10 repetitions, 3 sessions a week for 4 weeks.

SUMMARY:
the study was conducted to find out the effects of scapulothoracic joint mobilization with or without acromioclavicular joint mobilization in patients with sub-acromial pain syndrome.

DETAILED DESCRIPTION:
the study was conducted to determine the effects on the pain, range of motion of shoulder joint and the SPADI score in patients with sub-acromial pain syndrome post intervention including scapulothoracic upward rotation, posterior tilting and outward rotation glide with or without combination of acromioclavicular inferior glide.

ELIGIBILITY:
Inclusion Criteria: -Age 25 - 40 years

* Genders both male and female
* Patients having unilateral non-traumatic shoulder pain
* Patients having pain for ≥ 3 months
* According to Dutch Orthopedic Association Clinical Practice Guidelines 2 out of following 3 tests should be positive i.e. Hawkin's kennedy test, Painful arc test, and Infraspinatus resistance test
* Positive scapular assistance test
* Positive AC joint scarf test

Exclusion Criteria: - Patients having bilateral shoulder pain

* Younger than 25 and older than 40 years
* With positive drop arm test for supraspinatus tears
* Degenerative joint disease of shoulder
* Patients diagnosed with frozen shoulder
* Having history of shoulder fracture and dislocation
* Patients diagnosed with cervical radiculopathy (19)
* Having history of shoulder or neck surgery (19)
* Patients who had steroid injections in shoulder joint in the past 6 months
* Patients having other neurological, orthopedic and systemic problems affecting the shoulder, neck and back

Exclusion Criteria:

-

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating scale | from enrolment to the end of 4 weeks of treatment
  this scale is used to evaluate pain. it consists of 11 points from 0 to 10, where 0 represents no pain, 1-3 represents mild pain, 4-6 moderate pain and 7-10 represents severe pain.
Shoulder Pain and Disability Index SPADI | from enrolment to the end of 4 weeks treatment
  this questionnaire consisting of 13 items is used to assess the severity of pain and difficulty while performing daily life activities. two subscales for pain and disability. uses a visual Analog scale or Numeric rating scale for each item, resulting in scores from 0-100 for each sub-scale, with higher scores indicating more pain or disability.

SECONDARY OUTCOMES:
goniometer for shoulder flexion ROM | from enrolment to the end of 4 weeks treatment
  changes in shoulder flexion range of motion was measured at baseline and after 4 weeks of treatment sessions using goniometer
Goniometer for shoulder extension ROM | from enrolment to the end of 4 weeks of treatment
  changes in the shoulder extension range of motion were measured at baseline and at the end of 4 weeks of treatment sessions using goniometer
Goniometer for shoulder abduction ROM | from enrolment to the end of 4 weeks treatment sessions
  changes in the shoulder abduction range of motion were measured at baseline and at the end of 4 weeks of treatment sessions by using goniometer
Goniometer for shoulder adduction ROM | from enrolment to the end of 4 weeks of treatment
  changes in shoulder adduction range of motion were measured at baseline and at the end of 4 weeks treatment sessions by using goniometer
Goniometer for shoulder external rotation ROM | from enrolment to the end of 4 weeks of treatment
  changes in shoulder external rotation range of motion were measured at baseline and at the end of 4 weeks of treatment sessions by using goniometer
goniometer for shoulder internal rotation ROM | from enrolment to the end of 4 weeks treatment
  changes in the shoulder internal rotation range of motion were measured at baseline and at the end of 4 weeks of treatment sessions by using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafiq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Dr.Sheharyar Tanveer Clinic Sharaq pur, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Miguel Valtierra L, Salom Moreno J, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL. Ultrasound-Guided Application of Percutaneous Electrolysis as an Adjunct to Exercise and Manual Therapy for Subacromial Pain Syndrome: A Randomized Clinical Trial. J Pain. 2018 Oct;19(10):1201-1210. doi: 10.1016/j.jpain.2018.04.017. Epub 2018 May 16. PMID 29777953
- [Background] Park SJ, Kim SH, Kim SH. Effects of Thoracic Mobilization and Extension Exercise on Thoracic Alignment and Shoulder Function in Patients with Subacromial Impingement Syndrome: A Randomized Controlled Pilot Study. Healthcare (Basel). 2020 Sep 2;8(3):316. doi: 10.3390/healthcare8030316. PMID 32887287
- [Background] Ekici G, Özcan Ş, Öztürk BY, Öztürk B, Ekici B. Effects of deep friction massage and dry needling therapy on night pain and shoulder internal rotation in subacromial pain syndrome: 1-year follow up of a randomised controlled trial. International Journal of Therapy And Rehabilitation. 2021;28(2):1-12.
- [Background] Sharma S, Ejaz Hussain M, Sharma S. Effects of exercise therapy plus manual therapy on muscle activity, latency timing and SPADI score in shoulder impingement syndrome. Complement Ther Clin Pract. 2021 Aug;44:101390. doi: 10.1016/j.ctcp.2021.101390. Epub 2021 Apr 19. PMID 33901859
- [Background] Sharma S, Ghrouz AK, Hussain ME, Sharma S, Aldabbas M, Ansari S. Progressive Resistance Exercises plus Manual Therapy Is Effective in Improving Isometric Strength in Overhead Athletes with Shoulder Impingement Syndrome: A Randomized Controlled Trial. Biomed Res Int. 2021 Jun 30;2021:9945775. doi: 10.1155/2021/9945775. eCollection 2021. PMID 34307681
- [Background] Dunning J, Butts R, Fernandez-de-Las-Penas C, Walsh S, Goult C, Gillett B, Arias-Buria JL, Garcia J, Young IA. Spinal Manipulation and Electrical Dry Needling in Patients With Subacromial Pain Syndrome: A Multicenter Randomized Clinical Trial. J Orthop Sports Phys Ther. 2021 Feb;51(2):72-81. doi: 10.2519/jospt.2021.9785. Epub 2020 Aug 28. PMID 32857944
- [Background] Lyng KD, Andersen JD, Jensen SL, Olesen JL, Arendt-Nielsen L, Madsen NK, Petersen KK. The influence of exercise on clinical pain and pain mechanisms in patients with subacromial pain syndrome. Eur J Pain. 2022 Oct;26(9):1882-1895. doi: 10.1002/ejp.2010. Epub 2022 Jul 27. PMID 35852027
- [Background] Mohammed AH, Mahmoud NA, Abd El-Naeem MA, Abd El-Azeim AS. Efficacy of the Mulligan technique on subacromial space in patients with shoulder impingement syndrome. Physiotherapy Quarterly. 2024;32(3).
- [Background] Celik EB, Tuncer A. Comparing the Efficacy of Manual Therapy and Exercise to Synchronized Telerehabilitation with Self-Manual Therapy and Exercise in Treating Subacromial Pain Syndrome: A Randomized Controlled Trial. Healthcare (Basel). 2024 May 24;12(11):1074. doi: 10.3390/healthcare12111074. PMID 38891149
- [Background] Tauqeer S, Arooj A, Shakeel H. Effects of manual therapy in addition to stretching and strengthening exercises to improve scapular range of motion, functional capacity and pain in patients with shoulder impingement syndrome: a randomized controlled trial. BMC Musculoskelet Disord. 2024 Mar 2;25(1):192. doi: 10.1186/s12891-024-07294-4. PMID 38431547